CLINICAL TRIAL: NCT06094361
Title: "IONTOPHORESIS vs. PHONOPHORESIS": WHICH IS A BEST WAY TO TREAT SUBACROMIAL IMPINGEMENT SYNDROME? A RANDOMIZED STUDY
Brief Title: "IONTOPHORESIS vs. PHONOPHORESIS" for Treatment of Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Research Assisstant, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02.06.2015.284
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Iontophoresis; Phonophoresis; Pain; Disability
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain | interventions — Phonophoresis

STUDY DESIGN:
Intervention Model Description: There were two separate groups in the study. The first group received iontophoresis and the other group received phonophoresis. The effects on treatment outcomes were compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IONTOPHORESIS (Experimental): The group that received 75 mg diclofenac sodium with Chattanooga Physio device.
  Interventions: Procedure: Iontophoresis Intervention; Procedure: Conventional Therapy
- PHONOPHORESIS (Experimental): It is a treatment performed by applying 75 mg of 1% diclofenac sodium gel to the intervention area with the Chattanooga ultrasound device.
  Interventions: Procedure: Phonophoresis; Procedure: Conventional Therapy

INTERVENTIONS:
Procedure: Iontophoresis Intervention — Iontophoresis was applied with a Chattanooga Physio (DJO Global, Herentals, Belgium) brand device. The galvanic current mode was selected for the intervention. Intervention area was cleaned to prevent irritation and active electrode pad (cathode-5 cm2) was immersed in 75 mg diclofenac sodium solution. The current intensity of the application for 10 minutes was 0.1-0.2 mA/cm2.
  Arms: IONTOPHORESIS
Procedure: Phonophoresis — Phonophoresis was performed with a Chattanooga brand ultrasound device (Chattanooga, Intelect Legend Ultrasound, TN, USA). 75 mg gel containing 1% diclofenac sodium was applied to the shoulder area. The ultrasound was conducted continuously for 6 minutes with frequency of 1 MHz and an intensity of 1.5 watts/cm2.
  Arms: PHONOPHORESIS
Procedure: Conventional Therapy — All groups received a treatment program consisting of hot pack, Transcutaneous Electrical Nerve Stimulation and Shoulder girdle exercises for 30 minutes.

SUMMARY:
The aim of this study was to compare the effects of iontophoresis and phonophoresis applications added to conventional treatment on pain, range of motion, disability, and functional status in the shoulder region in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
Randomization: Forty-seven patients were assessed, and 43 completed the study in this randomized trial. The participants were divided into two groups (Iontophoresis:22 and Phonophoresis:21) using the online randomization software (www.randomizer.org). All patients gave written informed consent after being verbally informed about the study.

Assessment Period: Assessments were conducted twice, at the start and after completion of the 10-session treatment program.

Session Period: All treatment programs were delivered five days per week for two weeks. The total number of sessions was ten.

Analysis: The statistical analysis was performed using version 21 of the Statistical Package for the Social Sciences (SPSS).To verify normal distribution, the Shapiro-Wilk test and histogram curves were utilized. Descriptive statistics for parametric variables included mean, standard deviation, and percentage. Since the data exhibited normal distribution, independent sample T-tests were used for group comparison while paired sample T-tests were used to detect changes within the group. The significance level of p<0.05 was deemed acceptable for all analyses. For variables with nominal assessments, data were analyzed utilizing Yates Continuity Correction and Fisher's exact chi-square test.

The post hoc power of the study was calculated using Gpower 3.1.9.1 software. The resting VAS scores was taken as reference. In this context, Cohen's effect size was calculated as 1.00. When the alpha error was accepted as 5%, and effect size was 1.00, the post hoc power was found to be 94.27%.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Stage I-II SIS
* The ages between 18 and 65 years

Exclusion Criteria:

* Having underwent shoulder surgery,
* Participated in a shoulder-related treatment program within the previous six months,
* Failed to adhere to the treatment program by 70% or more

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | At the baseline
  This scale assess the pain of the patients. The scale is scored from 0-10, with 0 indicating no pain and 10 indicating intolerable pain.
Visual Analog Scale | Immediately after 10 physiotherapy sessions on consecutive days
  This scale assess the pain of the patients. The scale is scored from 0-10, with 0 indicating no pain and 10 indicating intolerable pain.

SECONDARY OUTCOMES:
Sociodemographic Data Form | At the baseline
  It is a form containing the descriptive characteristics of the patients.
Range of Motion | At the baseline
  The angular values of flexion, extension, abduction, internal and external rotation performed actively by the patients were examined with a universal goniometer.
Range of Motion | Immediately after 10 physiotherapy sessions on consecutive days
  The angular values of flexion, extension, abduction, internal and external rotation performed actively by the patients were examined with a universal goniometer.
Shoulder Disability Questionnaire | At the baseline
  This scale is a sixteen-item scale that assesses disability in individuals with shoulder complaints
Shoulder Disability Questionnaire | Immediately after 10 physiotherapy sessions on consecutive days
  This scale is a sixteen-item scale that assesses disability in individuals with shoulder complaints
Quick-Disabilities of the Arm, Shoulder and Hand Questionnaire | At the baseline
  In the scale, the functional status of individuals with shoulder pathology is questioned during their daily activities, and it is an assessment form filled by the patients themselves.
Quick-Disabilities of the Arm, Shoulder and Hand Questionnaire | Immediately after 10 physiotherapy sessions on consecutive days
  In the scale, the functional status of individuals with shoulder pathology is questioned during their daily activities, and it is an assessment form filled by the patients themselves.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No